CLINICAL TRIAL: NCT07188766
Title: Fluid Management in Sickle Cell Disease Vaso-occlusive Crisis: Restrictive Versus Liberal Strategies: A Randomized Controlled Trial (FLASC Trial)
Brief Title: Efficacy of Liberal Versus Restricted IV Fluid Approach in the Management of Sickle Cell Vaso-Occlusive Crisis
Acronym: FLASC
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Principal Investigator, Mohammed Saeed Saad Alshahrani, Consultant, Emergency and Critical Care Departments, Imam Abdulrahman Bin Faisal University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-01-0451
Record Dates: First submitted 2025-08-11; First posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: SCD; Vaso Occlussive Crisis
Keywords: sickle cell disease; sickle cell crisis; intravenous fluid; emergency department
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises; Emergencies | interventions — Sodium Chloride

STUDY DESIGN:
Intervention Model Description: This is a prospective, non-inferiority, open label multicenter randomized controlled trial. Patients on Intervention Group (Restricted approach group) will receive maintenance intravenous fluids at a keep-vein-open (KVO) rate and no extra intravenous fluids is administered.
  Control Group (Liberal Approach Group) Patients will receive an IV bolus of 20 mL/kg of normal saline or lactated Ringer's over 1 hour, followed by maintenance fluids at 1.5-2 ml/kg times the calculated daily maintenance requirements.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Restricted approach group (Experimental): Patients in this arm will receive maintenance intravenous fluids at a keep-vein-open (KVO) rate and no extra intravenous fluids is administered
  Interventions: Drug: Sodium Chloride (NaCl) 0.9 %
- Liberal Approach Group (Active Comparator): Patients will receive an IV bolus of 20 mL/kg of normal saline or lactated Ringer's over 1 hour, followed by maintenance fluids at 1.5-2 ml/kg times the calculated daily maintenance requirements
  Interventions: Drug: Sodium Chloride (NaCl) 0.9 %

INTERVENTIONS:
Drug: Sodium Chloride (NaCl) 0.9 % — Keep vein open rate
  Other Names: Restricted
  Arms: Restricted approach group
Drug: Sodium Chloride (NaCl) 0.9 % — IV bolus of 20 mL/kg of normal saline over 1 hour, followed by maintenance fluids at 1.5-2 ml/kg times the calculated daily maintenance requirements
  Other Names: Liberal
  Arms: Liberal Approach Group

SUMMARY:
Sickle cell disease (SCD) is a prevalent inherited blood disorder characterized by vaso-occlusive crises (VOCs), which lead to severe pain and complications. Despite hydration being a cornerstone of VOC management, the optimal fluid strategy remains uncertain. This study evaluates restrictive versus liberal fluid management strategies in patients with acute VOC.

This multi-center, open-label, non-inferiority RCT will enroll patients with SCD presenting with acute VOC. Participants will be randomized to either a restrictive or liberal intravenous fluid management protocol. Primary outcome is pain score reduction. Secondary outcomes include time to pain resolution, ED length of stay, hospital admission rate, cumulative opioid dose, adverse events (incidence of fluid overload, pulmonary congestion), acute chest syndrome, incidence of acute kidney injury, revisit rates within 72 hours of ED discharge, need for intensive care or high-dependency unit admission, need for additional interventions, and 28 days overall mortality. Data will be analyzed using intention-to-treat principles.

We hypothesize that a restrictive fluid strategy will achieve non-inferior pain control compared to a liberal strategy, while minimizing fluid-related complications. This study will provide evidence to inform clinical guidelines for fluid management in SCD patients experiencing VOCs.

DETAILED DESCRIPTION:
This study is a prospective, non-inferiority, open-label, multicenter randomized-controlled trial (RCT) conducted in the emergency departments (EDs) of tertiary care hospitals in Saudi Arabia. The primary objective is to compare two fluid management strategies- restrictive (intervention) vs. liberal (control) in adult sickle cell disease (SCD) patients hospitalized for VOC. The study evaluates whether a restrictive fluid approach is non-inferior to a liberal strategy in terms of pain resolution, hospitalization duration, and other clinical outcomes.

Patients will be randomized upon ED admission, and their assigned fluid regimen will be administered within the first hour. Clinical teams will monitor outcomes throughout hospitalization or up to 28 days post-enrollment.

Study Population

1. Recruitment Screening: All patients admitted to the ED with VOC will be screened for eligibility.

   Consent Model: A priori informed written consent will be obtained from conscious, coherent patients or substitute decision-makers.
2. Inclusion Criteria Age >18 years with confirmed SCD diagnosis.

   Presenting with VOC requiring hospitalization.

   Willingness to participate and provide informed consent.
3. Exclusion Criteria Requiring specialized IVF management per physician discretion.

Cardiac/Renal Conditions:

Congestive heart failure (CHF) or symptomatic systolic heart failure.

Chronic kidney disease (CKD), acute kidney injury (AKI), or renal transplantation.

Hemodynamic Instability:

Shock (SBP <100 mmHg or MAP <65) with hypoperfusion signs.

Other Exclusions:

Known/suspected pregnancy.

Prior enrollment in this trial within the last 30 days.

Concurrent enrollment in another trial affecting fluid management.

Inability to obtain IV access.

Trial Intervention

1. Screening & Randomization Screening occurs upon ED admission; evaluations must precede randomization.

   A screening log will track eligible vs. randomized patients.
2. Informed Consent A-priori consent model used due to the conscious-coherent state of most SCD patients in VOC.

   Efforts will be made to obtain consent immediately from the patient or surrogate.
3. Intervention Arms A. Intervention (Restrictive)Keep-vein-open (KVO) rate only (minimal fluids to maintain IV patency). No additional IV fluids administered.

B. Control (Liberal) 20 mL/kg IV bolus (NS or LR over 1 hour) + maintenance fluids (1.5-2 mL/kg/day).

Initiation: Both regimens start within 1 hour of ED admission and continue until ED discharge.

Hospitalized Patients:

Pain scores (NPRS) recorded at 24 & 48 hours. Total fluid intake documented at hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 years old with a confirmed diagnosis of SCD.
2. Presenting with a VOC.
3. Willingness to participate and provide informed consent.

Exclusion Criteria:

1. Patient requiring specialized IVF management as per the treating physician discretion.
2. Patients with congestive heart failure, and /or acute or chronic symptomatic systolic heart failure
3. Patients with a history of chronic kidney disease, acute kidney injury or renal transplantation
4. Patients with signs of shock (low SBP <100 or MAP < 65) and signs of hypo perfusion
5. Known or suspected pregnancy
6. Previously enrolled in this trial within the last 30 days
7. Enrolled in another trial study that interfered with fluid management
8. Unable to obtain IV access.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 394 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Change in Pain intensity | Baseline (within 30 minutes post admission), 1 hour, then hourly until ED discharge or 24- and 48-hours post-admission ( for admitted patients)
  Measured using the Numeric Pain Rating Scale (NPRS)

SECONDARY OUTCOMES:
Time to pain resolution | up to 4 hours
  NPRS score of ≤5
ED length of stay | at least 4 hours
  time elapsed from ED admission to ED discharge or admit to the wards
Hospital admission rate | within 24 hours of ED admission
  Proportion of participants requiring inpatient admission
Cumulative Opioid Dose | up to 4 hours
  Total opioid consumption during acute VOC episode
Revisit Rates | within 72 hours post ED discharge
  Percentage of patients who revisited the emergency department
Overall Mortality | within 28 days post-enrollment
  number of patients who died
Adverse events | up to 7 days
  total number of patients who encountered allergic reactions, respiratory distress, pulmonary edema, and acute chest syndrome, development of tachypnea, hypoxia, cough, crackles on auscultation, elevated BP, need for respiratory support, heart failure (worsening of tachycardia, hepatomegaly, peripheral edema, and allergic reactions (urticaria, angioedema, hypotension, wheezing)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed S Alshahrani, MD, Principal Investigator — King Fahd Hospital of the University- Imam Abdulrahman Bin Faisal University

IPD SHARING:
Plan to Share IPD: Yes
1. Demographics: Age, sex, and other baseline characteristics.
  2. Outcome Measures: primary and secondary outcomes of the trial.
  3. Adverse Events: Data on side effects or other adverse events participants experienced during the trial.
  4. Treatment Allocations: Information on which participants were assigned to each treatment group.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Background] Puri L, Nottage KA, Hankins JS, Anghelescu DL. State of the Art Management of Acute Vaso-occlusive Pain in Sickle Cell Disease. Paediatr Drugs. 2018 Feb;20(1):29-42. doi: 10.1007/s40272-017-0263-z. PMID 28853040
- [Background] Rizio AA, Bhor M, Lin X, McCausland KL, White MK, Paulose J, Nandal S, Halloway RI, Bronte-Hall L. The relationship between frequency and severity of vaso-occlusive crises and health-related quality of life and work productivity in adults with sickle cell disease. Qual Life Res. 2020 Jun;29(6):1533-1547. doi: 10.1007/s11136-019-02412-5. Epub 2020 Jan 13. PMID 31933113
- [Background] Okomo U, Meremikwu MM. Fluid replacement therapy for acute episodes of pain in people with sickle cell disease. Cochrane Database Syst Rev. 2015 Mar 12;(3):CD005406. doi: 10.1002/14651858.CD005406.pub4. PMID 25764071
- [Background] Brandow AM, Carroll CP, Creary S, Edwards-Elliott R, Glassberg J, Hurley RW, Kutlar A, Seisa M, Stinson J, Strouse JJ, Yusuf F, Zempsky W, Lang E. American Society of Hematology 2020 guidelines for sickle cell disease: management of acute and chronic pain. Blood Adv. 2020 Jun 23;4(12):2656-2701. doi: 10.1182/bloodadvances.2020001851. PMID 32559294
- [Background] Rosa RM, Bierer BE, Thomas R, Stoff JS, Kruskall M, Robinson S, Bunn HF, Epstein FH. A study of induced hyponatremia in the prevention and treatment of sickle-cell crisis. N Engl J Med. 1980 Nov 13;303(20):1138-43. doi: 10.1056/NEJM198011133032002. PMID 6999348
- [Background] GBD 2021 Sickle Cell Disease Collaborators. Global, regional, and national prevalence and mortality burden of sickle cell disease, 2000-2021: a systematic analysis from the Global Burden of Disease Study 2021. Lancet Haematol. 2023 Aug;10(8):e585-e599. doi: 10.1016/S2352-3026(23)00118-7. Epub 2023 Jun 15. PMID 37331373